CLINICAL TRIAL: NCT05890846
Title: Personalized Brain Functional Sectors (pBFS) Guided Transcranial Magnetic Stimulation (TMS) Treatment for Autism Spectrum Disorder (ASD): a Sham-controlled, Double-blinded, Randomized Clinical Trial Study
Brief Title: Precision TMS Treatment Guided by Personalized Brain Functional Sectors (pBFS) for ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Collaborators: Henan Provincial People's Hospital (Other); China Rehabilitation Research Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPASD2023DL
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder
Keywords: TMS; personalized medicine; ASD; fMRI
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DLPFC group (Experimental): Active iTBS will be delivered to the cognitive control network at left DLPFC.
  Interventions: Device: active iTBS; Behavioral: traditional 1on1 course
- Sham group (Sham Comparator): Sham iTBS will be delivered to the cognitive control network at left DLPFC.
  Interventions: Device: sham iTBS; Behavioral: traditional 1on1 course

INTERVENTIONS:
Device: active iTBS — Each participant will receive 1800 pulse active iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 12 weeks.
  Arms: DLPFC group
Device: sham iTBS — Each participant will receive 1800 pulse sham iTBS (100% RMT) in each session, 3 sessions per day, 5 days per week for 12 weeks.
  Arms: Sham group
Behavioral: traditional 1on1 course — Between every two iTBS sessions, the participant will receive a personalized 30-minutes one-on-one behavioral course, 2 courses per day, 5 days per week for 12 weeks.

SUMMARY:
This study will evaluate the efficacy and safety of pBFS-guided TMS treatment for the core symptom in autism spectrum disorder children, adolescents and young adults.

DETAILED DESCRIPTION:
Autism spectrum disorder is a neurodevelopmental disorder characterized by impaired social communication and repetitive behaviors. Broad cognitive control function deficit in ASD suggested cognitive control function as a potential phenotype and treatment target. Using the personalized Brain Functional Sectors (pBFS) technique, investigators could precisely identify individualized brain areas underlying cognitive control function based on the task free functional MRI data. The tailored TMS intervention target to cognitive control function network which located in the left dorsal lateral prefrontal cortex (DLPFC) will be selected for each participant by a blinded researcher.

The participants will be equally randomized to the active iTBS to the cognitive control function network, and sham iTBS at a ratio of 2:1. Each participant will receive 5 days of treatment per week for 12 weeks. Functional MRI data under sedation will be collected pre-and post-treatment. Three behavioral evaluations will be taken pre-treatment, after 8-weeks treatment and after 12-weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Nearest age 6-30 years old
* Have the diagnosis of autism spectrum disorder
* ADOS-2 score is higher than the ASD cut-offs
* Capacity to follow the study procedures, including fMRI scan under sedation, assessment, and rehabilitation training
* Participant's parent or other legal guardian give informed consent

Exclusion Criteria:

* Current or history of psychotic disorders, such as schizophrenia, schizoaffective disorder, bipolar disorder
* Severe self-injury or suicidal behavior presented in the last one year
* Severe visual, auditory, or motor disability that interferes with any study procedure
* Current or history of seizure
* Known severe physical diseases, such as congenital heart defect, traumatic brain injury
* Metal implantations, which are contradicted by MRI or TMS, such as artificial cardiac pacemakers, stents, cochlear implants
* Received TMS, tCS, FUS, or other neuromodulation treatment in the last 3 months
* Currently participating in other clinical trials

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Response rate after 12 weeks treatment | Pre-treatment (baseline), after 12-weeks treatment
  Treatment response is defined as improvement, i.e., scores decreased, in both the social affect (SA) dimension score change of autism diagnostic observation scale, 2nd edition (ADOS-2) from baseline. For ADOS-2 SA, higher scores means more severe symptom.

SECONDARY OUTCOMES:
Response rate after 8 weeks treatment | Pre-treatment (baseline), after 8-weeks treatment
  Treatment response is defined as improvement, i.e., scores decreased, in the social affect (SA) dimension score change of autism diagnostic observation scale, 2nd edition (ADOS-2) from baseline. For ADOS-2 SA, higher scores means more severe symptom.
ADOS-2 SA score change | Pre-treatment (baseline), after 8-weeks treatment，after 12-weeks tretment
  The ADOS-2 SA score changes from baseline. Higher scores mean a worse outcome.
SCQ score change | Pre-treatment (baseline), after 8-weeks treatment，after 12-weeks tretment
  SCQ score change from baseline. Higher scores mean a worse outcome.
ADOS-2 total score change | Pre-treatment (baseline), after 8-weeks treatment，after 12-weeks tretment
  The ADOS-2 total score change from baseline. Higher scores mean a worse outcome.
CBCL score change | Pre-treatment (baseline), after 8-weeks treatment，after 12-weeks tretment
  Score change of the child behavior checklist (CBCL) from baseline. Higher scores mean a worse outcome.
SRS-2 score change | Pre-treatment (baseline), after 8-weeks treatment，after 12-weeks tretment
  Score change of the Social Responsiveness Scale, 2nd edition (SRS-2) from baseline. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (2):
- China (2):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - China Rehabilitation Research Center, Beijing